CLINICAL TRIAL: NCT03270423
Title: PathMate2: The Impact of Health Information System Services on the Effects of Therapy in Overweight Teenagers
Acronym: PM2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ostschweizer Kinderspital (Other)
Responsible Party: Principal Investigator, Dagmar l'Allemand, Prof. Dr. med., Ostschweizer Kinderspital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-01965
Record Dates: First submitted 2017-07-26; First posted 2017-09-01 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Obesity, Adolescent
MeSH Terms: conditions — Pediatric Obesity | interventions — Infection Control, Dental

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention SG (Active Comparator): Therapy during 6 months with PathMate2 design. 6 therapy visits + PathMate2 over 6 months
  Interventions: Device: PathMate2
- Control SG (No Intervention): Therapy during 6 months with usual care. 10 therapy visits over 6 months
- Intervention VD (Active Comparator): Adapted sport session 1h/week + PathMate-S during 6 months
  Interventions: Device: PathMateS
- Control VD (No Intervention): Adapted sport session 1h/week during 6 months

INTERVENTIONS:
Device: PathMate2 — To improve self-regulation of overweight adolescents and subsequently their weight status, we tested, whether a biofeedback relaxation exercise decreases stress and whether relaxation services as well as sensor data integration implemented in a novel Smartphone App supported intervention have effects on stress, physical activity and weight outcomes. During the intensive phase of 6 months, patients of the intervention group (IG) are equipped with a smartphone and a specially designed chat App with game character, which encourages them through a virtual coach to achieve daily activity, healty lifestyle or relaxation challenges and earn virtual rewards, to increase adherance to the health information system.
  Other Names: Mobile-coach obesity intervention in adolescents
  Arms: Intervention SG
Device: PathMateS — Overweight or obese adolescents of the treatment as-usual group (CG) have monthly visits on site during the intensive phase. Counseling for physical activity, healthy eating and lifestyle as well as psychosocial wellbeing is provided by a pediatrician.
  Other Names: controls
  Arms: Intervention VD

SUMMARY:
Randomised controlled trial in overweight adolescents using a health App.

DETAILED DESCRIPTION:
Problem In Switzerland, 20% of children are overweight and novel methods are urgently needed to control the epidemic. Foundations of chronic diseases develop during childhood and track into adulthood obesity in more than 75% of patients, contributing to a significant increase in public health costs.

Multi-professional programs combining physical activity, nutritional and behavioral components have positive effects on therapy outcomes and co-morbidities, but these interventions induce high costs and are time-consuming for health providers, patients and families, in particular those living in rural regions. In fact, less than 0.2% of overweight children can participate in these programs. Thus, health information systems (HIS) have not only the potential to improve outcomes of obesity therapy but also to reduce health costs and increase access to health care in remote regions. Most HIS have indeed not been evaluated in this regard.

Preparation work In the PathMate project (SNF grant #135552), a mobile HIS has been developed for teenagers to support therapy and to prevent obesity in accordance with state-of-the-art multiprofessional programs and, in contrast to commercially available IT applications, with a high standard of data protection and safety. The IS effects of this HIS have been successfully evaluated in first longitudinal studies. In parallel, the impact of multi-professional therapies in Swiss children as well as potential confounders have been established in several longitudinal cohort studies with up to two-years follow-up.

Objectives

The overall goal of PathMate2 is to assess the impact of HIS services on the degree of obesity measured by the body mass index (BMI) incl. other health outcomes. Individual and shared understanding between patients and therapists are assessed as mediating factors. Specific goals are:

1. to assess the effects of a child-friendly IT-mediated low-threshold intervention under the supervision of primary care providers and obesity experts, compared to expensive on-site consultations in highly specialized pediatric obesity centers
2. to automatically capture and process obesity-related biosignals by smart sensors and use results for immediate feedback for the patients and medical providers based on permissions and communication patterns and
3. to design evidence-based selfregulation interventions for teenager in their everyday life by coupling Neuro Information Systems (NeuroIS) services with Smart Health Sensors (SHS).

Methods HIS services are collaboratively developed by design-science research and evaluated by medical experts, patients, IS researcher and computer scientists. First, HIS services from PathMate are enhanced with SHS enabling real-time data analytics on mobile devices and results can be seen by both therapists and patients. Second, a randomized controlled trial (RCT) is conducted by a physician in a specialized pediatric obesity center in St. Gall with the goal to evaluate the effects of the re-designed and improved HIS services on adherence to therapy of the patient and his parents as well as on BMI and other health outcomes; a second RCT is conducted in parallel to assess the effects of these services in a community setting in the French-speaking part of Switzerland.

Importance and impact Building on the preliminary results of the PathMate project it is expected that the improved HIS services that are going to be designed and evaluated in PathMate2 have the potential for a significant impact on individual health and the quality of healthcare systems in general.

ELIGIBILITY:
Inclusion Criteria:

* obesity, BMI > P. 97 (Jenni et al., 2011) or overweight, BMI >P.90, plus risk factors or co-morbidity
* ability and parent's permission to use pre-configured study smartphones handed out to the children
* readiness to use the personal smartphone number and to spend the sum allocated exclusively for the study SMS during the 6 months of intervention

Exclusion Criteria:

* major somatic or psychiatric disease without adequate treatment,
* weight-relevant medication (antiepileptic drugs, methylphenhydate and similar medication),
* inability or lack of parent's or caregivers' permission to use a study smartphone with a mobile phone contract,
* lack of informed consent from children and parents and
* undue consumption of the amount allocated for study SMS for non-study purposes,
* overuse of smartphone e.g. without night beak for at least 8 hours.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | 12 months
  Main outcome parameter is Body Mass Index, as BMI-SDS adjusted for gender & age. Group size of 4*20 was based on an expected decrease by -0.23±0.02 (SDS, Mean±SD) after 1 year, from initially 2.88±0.7.

SECONDARY OUTCOMES:
fitness / physical capability | 12 months
  Eurofit-test
fitness / physical activity | 12 months
  accelerometry
stress reduction, biological measure | 12 months
  Cortisol levels in blood
stress and arousal | 12 months
  Self-Assessment Manikin (SAM) Scale
reduction of chronic stress | 12 months
  Trierer Stress Inventar questionnaire (TICS)
stress and arousal, biophysical measure | 12 months
  skin conductance (Nexus 10)
well-being | 12 months
  KIDSCREEN
waist circumference | 12 months
  Waist-to-Height-ratio or SDS according to Fredricks 2005

CONTACTS AND LOCATIONS:
Overall Officials: Dagmar lAllemand, Prof. MD, Principal Investigator — Ostschweizer Kinderspital, St. Gallen, Switzerland
Locations (1):
- Ostschweizer Kinderspital, Sankt Gallen, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haug S, Kowatsch T, Castro RP, Filler A, Schaub MP. Efficacy of a web- and text messaging-based intervention to reduce problem drinking in young people: study protocol of a cluster-randomised controlled trial. BMC Public Health. 2014 Aug 7;14:809. doi: 10.1186/1471-2458-14-809. PMID 25099872
- [Derived] Metzendorf MI, Wieland LS, Richter B. Mobile health (m-health) smartphone interventions for adolescents and adults with overweight or obesity. Cochrane Database Syst Rev. 2024 Feb 20;2(2):CD013591. doi: 10.1002/14651858.CD013591.pub2. PMID 38375882